CLINICAL TRIAL: NCT03846388
Title: Prediction Of Reproductive Outcome in Assisted Conception Cycles in Women With Unexplained Infertility
Brief Title: Reproductive Outcome in Assisted Conception Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACC
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with unexplained infertility (Other)
  Interventions: Diagnostic Test: follicular stimulating hormone; Diagnostic Test: Anti-mullerian hormone; Radiation: Basal antral follicle count
- patients with tubal, male factor or polycystic ovary syndrome (Other)
  Interventions: Diagnostic Test: follicular stimulating hormone; Diagnostic Test: Anti-mullerian hormone; Radiation: Basal antral follicle count

INTERVENTIONS:
Diagnostic Test: follicular stimulating hormone — in the serum of our patients
Diagnostic Test: Anti-mullerian hormone — in the serum of our patients
Radiation: Basal antral follicle count — by ultrasound

SUMMARY:
Infertility is the failure to conceive after regular unprotected sexual intercourse for one year. Primary infertility refers woman who has never conceived, and secondary infertility to one who has had a previous pregnancy.The most frequent causes for infertility are ovulatory disorder or anovulation (27-30%) , tubal factor(20-22%), abnormal semen parameters(45-50%). Unexplained infertility refers to infertile couples in whom standard investigations, including tests of ovulation, tubal patency tests and semen analysis are normal. incidence 15-17% of infertile couples. New guidelines on infertility recommend that women with unexplained infertility should be advised for expectant management for 2 years .If pregnancy is not achieved after this period In vitro fertilization Should be considered. The Fast Track and Standard Treatment trial demonstrated A shorter time to pregnancy and higher per cycle pregnancy rates for In vitro fertilization compared with treatment with oral agents or gonadotropins in Patients with unexplained infertility. Successful pregnancy after assisted reproductive technology is influenced by numerous predictors that have been investigated in the previous years. The central predictors of success are the sperm, oocyte quality and endometrial receptivity. Oocyte quality depends mainly on the age of the woman , and her ovarian reserve. Parameters most commonly studied are the woman's age , her antral follicle count , and laboratory tests including serum randomly done during the menstrual cycle levels at day 3 of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* in vitro fertilization treatment due to many factors including tubal, male, and unexplained factors.
* body mass index (BMI) (18-35)kg/m2

Exclusion Criteria

1. patient age less than 20 and more than 40 years.
2. body mass index less than 18 and more than 35 kg/m2.
3. period of infertility less than 2 years..
4. untreated hyperthyroidism, hypothyroidism, diabetes, hypertension.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
live birth rate | 12 months

SECONDARY OUTCOMES:
Number of fertilized oocytes | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided